CLINICAL TRIAL: NCT00296816
Title: A Pilot Phase II Study Evaluating the Combination of Oxaliplatin and Docetaxel With Bevacizumab as First Line Therapy in Patients With FIGO Stage IB-IV Epithelial Ovarian, Primary Peritoneal or Fallopian Tube Carcinoma
Brief Title: TEACO: Taxotere, Eloxatin, Avastin in Cancer of the Ovary
Acronym: TEACO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM_L_0239
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Docetaxel; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxaliplatin/Docetaxel/Bevacizumab (Experimental): Participants with International Federation of Gynecology and Obstetrics (FIGO) stage IB through IV ovarian, primary peritoneal, or fallopian tube carcinoma treated with Oxaliplatin, Docetaxel, and Bevacizumab - 28 days after initial surgery
  Interventions: Drug: Bevacizumab (Avastin®); Drug: Docetaxel (Taxotere®); Drug: Oxaliplatin (Eloxatin®)

INTERVENTIONS:
Drug: Bevacizumab (Avastin®) — 15 mg/kg bevacizumab administered intravenously (IV) over 30 to 90 minutes on Day 1 of every 3 week cycle for 12 months or until disease progression or unacceptable toxicity
Drug: Docetaxel (Taxotere®) — 75 mg/m^2 docetaxel was administered IV over 1 hour on Day 1 of every 3 week cycle for 6 cycles or until disease progression or unacceptable toxicity
Drug: Oxaliplatin (Eloxatin®) — 85 mg/m^2 Oxaliplatin was administered IV over 2 hours on Day 1 of every 3 week cycle for 6 cycles or until disease progression or unacceptable toxicity

SUMMARY:
Feasibility study to assess a novel combination of cytotoxic agents, docetaxel and oxaliplatin, as first-line therapy in the treatment of ovarian cancer and the impact of angiogenesis inhibition for the progression and prognosis of ovarian cancer by concurrent addition of bevacizumab (Avastin®).

DETAILED DESCRIPTION:
Participants were

* administered study medication approximately 28 days after initial surgery for ovarian cancer
* received the study treatment regimen of up to one year unless there was disease progression, unacceptable toxicity, death, participant refusal, or treatment delay beyond the time frame permitted for each treatment

Participants were followed for survival for a minimum 3 years from the date of enrollment

ELIGIBILITY:
INCLUSION CRITERIA:

1. Females 18 years of age or older
2. Participants with a histologic diagnosis of ovarian, primary peritoneal, or fallopian tube carcinoma, Stage Ib- IV, with either optimal (≤ 1 cm residual disease) or suboptimal residual disease ( > 1 cm maximal diameter any remaining lesion) following initial surgery.
3. Participants with the following histologic epithelial cell types are eligible: Serious adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma,undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma N.O.S.
4. Participant must have adequate bone marrow function
5. Participant must have adequate renal function
6. Participant must have adequate urine protein/creatinine reaction (UPC) of <1.0;
7. Participant must have adequate neurologic function
8. Hepatic function: Total Bilirubin ≤ ULN; AST and ALT and Alkaline Phosphatase must be within the range allowing for eligibility. In determining eligibility the more abnormal of the two values (AST or ALT) should be used.
9. Blood Coagulation parameters: PT such that international normalized ratio (INR) is < 1.5 (or an in-range INR, usually between 2 and 3, if a participant is on stable dose of therapeutic Warfarin or low molecular weight heparin) and a PTT < 1.2 times the upper limit normal.
10. Participants must be enrolled in the study prior to 50 days (every effort will be made for prior to 28 days) after initial surgery performed for the combined purpose of diagnosis, staging and cytoreduction.
11. Participants with measurable and non-measurable disease are eligible. Participants with suboptimal disease are eligible. Participants may or may not have cancer-related symptoms.
12. Participants who have met the pre-entry requirements specified including serologic measurement of CA-125 as a baseline for subsequent determination of response using Rustin criteria.
13. Participants with a GOG Performance Status of 0, 1, or 2.

EXCLUSION CRITERIA:

1. Participants with a current diagnosis of epithelial ovarian tumor of low malignant potential (Borderline carcinomas) are not eligible. Participants with a prior diagnosis of a low malignant potential tumor that was surgically resected and who subsequently develop invasive adenocarcinoma are eligible, provided that they have not received prior chemotherapy for any ovarian tumor.
2. Germ cell tumors, sex cord-stromal tumors, carcinosarcomas, mixed mullerian tumors or carcinosarcomas, metastatic carcinomas from other sites to the ovary and low malignant potential tumors including so called micropapillary serous carcinomas are not eligible.
3. Participants who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded. Prior radiation for localized cancer of the skin is permitted, provided that it was completed more than 5 years prior to enrollment, and the participant remains free of recurrent or metastatic disease.
4. Participants who have received any prior anticancer chemotherapy or biologic therapy for any malignancy are excluded.
5. Participants with synchronous primary endometrial cancer, or a past history of primary endometrial cancer, are excluded, unless all of the following conditions are met: Stage not greater than I-B; Less than 3 mm invasion without vascular or lymphatic invasion; No poorly differentiated subtypes, including papillary serous, clear cell, or other FIGO Grade 3 lesions.
6. Participants with any history of cancer, with the exception of inclusion criteria #2 and #3, and non-melanoma skin cancer, who are cancer free for the last 5 years, are excluded.
7. Participant with acute hepatitis or active infection that requires parenteral antibiotics.
8. Participants with serious, non-healing wound, ulcer, or bone fracture. This includes history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days.

   Participants with granulating incisions healing by secondary intention with no evidence of fascial dehiscence or infection are eligible but require weekly wound examinations.
9. Participants with active bleeding or pathologic conditions that carry high risk of bleeding,such as known bleeding disorder, coagulopathy, or tumor involving major vessels.
10. Participants with history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study.
11. Participants with clinically significant cardiovascular disease.
12. Participants with clinically significant proteinuria. Urine protein should be screened by urinalysis. Participants discovered to have a urine protein: serum creatinine ratio greater than or equal to 1 should undergo a 24-hour urine collection, which must be an adequate collection and must demonstrate < 1000 mg protein/24 hr to allow participation in the study.
13. Participants with or with anticipation of invasive procedures.
14. Participants with GOG Performance Grade of 3 or 4.
15. Participants who are pregnant or nursing.
16. Participants with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies and hypersensitivity to polysorbate 80 or hypersensitivity to any of the study drugs and its ingredients.
17. Participants who participated in a study with any investigational product/device within the last 30 days.
18. Any medical condition that in the judgment of the investigator would jeopardize any participant safety or the study drug evaluation for efficacy and safety.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2006-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, BS, MT (ASCP), Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 152 participants were screened for the study. 20 were screen failures. 132 participants met eligibity criteria and were treated with study medication.
Period: Overall Study
Arm/Group | Oxaliplatin/Docetaxel/Bevacizumab
Started | 132
Completed | 58 (Completed study treatment for a minimum of three years)
Not Completed | 74
Not completed — Disease Progression | 37
Not completed — Adverse Event | 18
Not completed — Investigator/Participant request | 5
Not completed — Non-compliance | 1
Not completed — Missing for end of treatment | 4
Not completed — Progression based on CA-125 (biomarker) | 2
Not completed — Poor performance status | 1
Not completed — Relocation to Florida | 1
Not completed — Noncompliance/decision to discontinue | 1
Not completed — Urine protein/creatinine ratio delay | 1
Not completed — Neuropathy/patient preference | 1
Not completed — Proteinuria | 1
Not completed — ineligibility due to radiation treatment | 1

BASELINE CHARACTERISTICS:
Groups:
- Oxaliplatin/Docetaxel/Bevacizumab (Measurable Disease): Participants with International Federation of Gynecology and Obstetrics (FIGO) stage IB through IV ovarian, primary peritoneal, or fallopian tube carcinoma treated with Oxaliplatin, Docetaxel, and Bevacizumab - 28 days after initial surgery, with a measurable disease at baseline.
  Measurable disease was defined as having at least one lesion that could be accurately measured in at least one dimension.
- Oxaliplatin/Docetaxel/Bevacizumab (Non-Measurable Disease): Participants with International Federation of Gynecology and Obstetrics (FIGO) stage IB through IV ovarian, primary peritoneal, or fallopian tube carcinoma treated with Oxaliplatin, Docetaxel, and Bevacizumab - 28 days after initial surgery, who did not have a measurable disease at baseline.
  Measurable disease was defined as having at least one lesion that could be accurately measured in at least one dimension.
- Total: Total of all reporting groups
Arm/Group | Oxaliplatin/Docetaxel/Bevacizumab (Measurable Disease) | Oxaliplatin/Docetaxel/Bevacizumab (Non-Measurable Disease) | Total
Number analyzed (Participants) | 80 | 52 | 132
Age Continuous [Mean (Standard Deviation); unit: years] | 57.5 (10.43) | 60.9 (9.54) | 58.8 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 52 | 132
  Male | 0 | 0 | 0
Primary Tumor Site [Number; unit: participants]
  Ovary | 65 | 45 | 110
  Fallopian tube | 6 | 5 | 11
  Peritoneum | 9 | 2 | 11
FIGO stage at diagnosis [Number; unit: participants] — Ovarian cancer staging at diagnosis was based on the International Federation of Gynecology and Obstetrics (FIGO).
  * Stage I is the least severe, where the tumor is restricted to the ovaries.
  * Stage II involves both ovaries and the pelvis.
  * Stage III involves the ovaries and has microscopically confirmed peritoneal metastasis outside the pelvis and/or regional lymph node (also includes liver capsule metastasis).
  * Stage IV involves distant metastasis beyond the peritoneal cavity.
  participants
    Stage IB | 0 | 0 | 0
    Stage IC | 0 | 3 | 3
    Stage IIA | 0 | 0 | 0
    Stage IIB | 0 | 0 | 0
    Stage IIC | 3 | 5 | 8
    Stage IIIA | 3 | 2 | 5
    Stage IIIB | 2 | 5 | 7
    Stage IIIC | 57 | 32 | 89
    Stage IV | 15 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Twelve-month Progression-free Survival (PFS) Rate in Participants
Description: Tumor assessments were performed by Computed tomography (CT) and Magnetic Resonance Imaging (MRI) to evaluate disease progression based on Gynecologic Oncology Group (GOG) Response Evaluation Criteria in Solid Tumors (RECIST).
  Disease progression was recorded as any one of the following:
  * appearance of a new lesion
  * symptomatic deterioration
  * progression of target or nontarget lesions
  * death
  Participants who did not die or show show disease progression achieved PFS. PFS rate is the percent of participants who achieved PFS.
Time Frame: up to 12 months following treatment initiation
Population: Intent-to-treat population with measurable disease at baseline - All participants with measurable disease at baseline who received study drugs, except for participants from one site which was closed prematurely, and for whom efficacy data was not available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oxaliplatin/Docetaxel/Bevacizumab
Number analyzed (Participants) | 70
percentage of participants | 65.7 [53.4 to 76.7]

2. Secondary Outcome: Twenty Four-month Progression-free Survival (PFS) Rate in Participants
Description: as for outcome 1
Time Frame: up to 24 months following treatment initiation
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oxaliplatin/Docetaxel/Bevacizumab
Number analyzed (Participants) | 70
percentage of participants | 34.3 [23.3 to 46.6]

3. Secondary Outcome: Median Time to Progression-free Survival (PFS)
Description: Time to PFS was the interval from the date of registration to the earliest date of disease progression or death, whichever occurred first.
  Time of PFS was censored
  * on the last available tumor assessment date for participants leaving the study prior to disease progression or death; and also for participants requiring off-study medication or additional debulking surgery (where assessment date used was the one prior to off-study medication or surgery),
  * at Day 1, for living participants with no post-baseline tumor assessments.
  Median PFS was estimated from a Kaplan-Meier curve.
Time Frame: up to approximately 1300 days following treatment initiation
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Oxaliplatin/Docetaxel/Bevacizumab
Number analyzed (Participants) | 70
days | 495 [384 to 596]

4. Secondary Outcome: Tumor Response Rate Based on Gynecologic Oncology Group (GOG) Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Tumors were assessed by CT and MRI. Tumor response was evaluated by GOG RECIST in which:
  * Complete response (CR) was the disappearance of all target and non-target lesions, with no evidence of new lesions
  * Partial response (PR) was at least a 30% decrease in the sum of longest dimensions (LD) of all measurable target lesions
  Participants with a response (CR or PR) were to have the initial response confirmed by tumor imaging in 4-6 weeks.
Time Frame: up to 12 months following treatment initiation
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Docetaxel/Bevacizumab
Number analyzed (Participants) | 70
participants
  Unconfirmed response (CR+PR) | 51
  Unconfirmed complete response (CR) | 23
  Unconfirmed partial response (PR) | 28
  Unconfirmed progressive disease (PD) | 5
  Confirmed response (CR+PR) | 41
  Confirmed complete response (CR) | 21
  Confirmed partial response (PR) | 20

5. Secondary Outcome: Twelve-month Recurrence-free Survival (RFS) Rate in Participants With Non Measurable Disease at Baseline
Description: Participants with Recurrence-free survival (RFS) were participants with a non-measurable disease at baseline, who had not achieved disease progression nor had died.
  Disease progression included the following:
  * the appearance of a new lesion
  * symptomatic deterioration
  * progression of non-target lesions
  * a predefined serum CA 125 increase.
  RFS rate was the percent of participants in the non-measurable disease subgroup who achieved RFS.
Time Frame: up to 12 months following treatment initiation
Population: All participants with non-measurable disease at baseline, except for those at one site that closed prematurely, as their data was not available for efficacy measures.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oxaliplatin/Docetaxel/Bevacizumab
Number analyzed (Participants) | 40
percentage of participants | 67.5 [50.9 to 81.4]

6. Secondary Outcome: Median Time to Recurrence-free Survival (RFS) in Participants With Non-measurable Disease at Baseline
Description: The time to RFS was programmatically defined as the interval from the date of registration to the earliest date of disease progression or death, whichever occurred first.
  Participants were
  * censored on the last available CA 125 biomarker blood draw date if
    * left the study prior to disease progression or death
    * they received off-study anti-tumor medication
    * underwent debulking surgery
  * censored at Day 1 if they were alive had no post baseline CA 125 biomarker blood draw.
Time Frame: up to approximately 1500 days following treatment initiation
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Oxaliplatin/Docetaxel/Bevacizumab
Number analyzed (Participants) | 40
days | 631 [427 to NA] — Some participants did not show recurrence and were living, therefore the upper limit is not applicable

7. Secondary Outcome: CA-125 Response Rate
Description: A CA-125 response was considered at least a 50% reduction in the level of the biomarker, CA-125, from a pretreatment level, which was confirmed and maintained for at least 28 days.
  The overall CA-125 biomarker response rate was defined as the number of participants in the measurable disease subgroup who met the above criteria at least once within the study treatment period +21 days, divided by the number of evaluable participants in the disease subgroup.
Time Frame: up to 12 months after treatment initiation
Population: All participants with non-measurable and measurable disease at baseline, and a pretreatment sample that was at least twice the ULN value for CA-125 within 2 weeks of first study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oxaliplatin/Docetaxel/Bevacizumab
Number analyzed (Participants) | 80
percentage of participants
  With non-measurable disease at baseline (N=27) | 81.5 [61.9 to 93.7]
  With measurable disease at baseline (N=53) | 83.0 [70.2 to 91.9]

8. Secondary Outcome: Overall Survival Rate
Description: Survival was the observed length of life from entry into the study to death or the date of last contact.
  The overall survival rate (percentage of participants showing survival) at 12 and 24-months is reported here.
Time Frame: up to up to approximately 1700 days after treatment initiation
Population: Intent-to-treat population - All participants who received study drugs, except for participants from one site which was closed prematurely, and for whom efficacy data was not available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oxaliplatin/Docetaxel/Bevacizumab
Number analyzed (Participants) | 110
percentage of participants
  Overall survival at 12 months | 85.5 [77.5 to 91.5]
  Overall survival at 24 months | 71.8 [62.4 to 80.0]

9. Secondary Outcome: Median Overall Survival Time
Description: Survival was the observed length of life from entry into the study to death or the date of last contact.
  The median overall survival time was estimated using Kaplan-Meier Curve.
Time Frame: up to approximately 1700 days after treatment initiation
Population: as for outcome 8
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Oxaliplatin/Docetaxel/Bevacizumab
Number analyzed (Participants) | 110
days | 1437.0 [1036.0 to NA] — Some participants were living, therefore the upper limit is not applicable

ADVERSE EVENTS:
Description: AEs were collected up to 30 days after the administration of the last study dose.
Arm/Group | Oxaliplatin/Docetaxel/Bevacizumab
Serious Adverse Events (participants affected / at risk) | 33/132
Other Adverse Events (participants affected / at risk) | 130/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin/Docetaxel/Bevacizumab (N=132)
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Small intestinal obstruction (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colonic fistula (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Peritoneal adhesions (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5
Hypertension (Vascular disorders) | 1
Poor venous access (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin/Docetaxel/Bevacizumab (N=132)
Neutropenia (Blood and lymphatic system disorders) | 59
Leukopenia (Blood and lymphatic system disorders) | 31
Anaemia (Blood and lymphatic system disorders) | 18
Lymphopenia (Blood and lymphatic system disorders) | 13
Lacrimation increased (Eye disorders) | 35
Vision blurred (Eye disorders) | 10
Nausea (Gastrointestinal disorders) | 85
Diarrhoea (Gastrointestinal disorders) | 77
Constipation (Gastrointestinal disorders) | 59
Vomiting (Gastrointestinal disorders) | 42
Abdominal pain (Gastrointestinal disorders) | 37
Stomatitis (Gastrointestinal disorders) | 26
Abdominal discomfort (Gastrointestinal disorders) | 11
Abdominal pain lower (Gastrointestinal disorders) | 10
Dysphagia (Gastrointestinal disorders) | 10
Gingival bleeding (Gastrointestinal disorders) | 10
Oral pain (Gastrointestinal disorders) | 10
Abdominal distension (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 8
Flatulence (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 101
Oedema peripheral (General disorders) | 19
Asthenia (General disorders) | 12
Pain (General disorders) | 12
Malaise (General disorders) | 11
Pyrexia (General disorders) | 10
Chest pain (General disorders) | 9
Mucosal inflammation (General disorders) | 9
Temperature intolerance (General disorders) | 9
Hypersensitivity (Immune system disorders) | 8
Urinary tract infection (Infections and infestations) | 30
Upper respiratory tract infection (Infections and infestations) | 14
Sinusitis (Infections and infestations) | 11
Rhinitis (Infections and infestations) | 10
Nasopharyngitis (Infections and infestations) | 7
Alanine aminotransferase increased (Investigations) | 12
Aspartate aminotransferase increased (Investigations) | 12
Neutrophil count (Investigations) | 12
Blood alkaline phosphatase increased (Investigations) | 10
Weight decreased (Investigations) | 7
Decreased appetite (Metabolism and nutrition disorders) | 44
Hypokalaemia (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 47
Back pain (Musculoskeletal and connective tissue disorders) | 26
Myalgia (Musculoskeletal and connective tissue disorders) | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7
Neuropathy peripheral (Nervous system disorders) | 64
Headache (Nervous system disorders) | 40
Peripheral sensory neuropathy (Nervous system disorders) | 33
Dysgeusia (Nervous system disorders) | 31
Paraesthesia (Nervous system disorders) | 26
Dizziness (Nervous system disorders) | 24
Hypoaesthesia (Nervous system disorders) | 8
Insomnia (Psychiatric disorders) | 20
Depression (Psychiatric disorders) | 19
Anxiety (Psychiatric disorders) | 9
Proteinuria (Renal and urinary disorders) | 11
Dysuria (Renal and urinary disorders) | 10
Vaginal haemorrhage (Reproductive system and breast disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 39
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10
Alopecia (Skin and subcutaneous tissue disorders) | 86
Nail disorder (Skin and subcutaneous tissue disorders) | 33
Rash (Skin and subcutaneous tissue disorders) | 17
Dry skin (Skin and subcutaneous tissue disorders) | 15
Nail discolouration (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 7
Hypertension (Vascular disorders) | 31
Flushing (Vascular disorders) | 14
Hot flush (Vascular disorders) | 10

LIMITATIONS AND CAVEATS:
One site closed prematurely during the study. Every effort was made to collect, at minimum, any outstanding safety data for the participants at this site. As a result, participants from this site were included only in the safety analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor encourages the publication of the results of their studies, using only clean, checked and validated data in order to ensure the accuracy of the results.

At least 45 days in advance of proposed submission, the Investigator should forward a copy of the manuscript or abstract for review by the sponsor, and, if necessary, delay publication or communication for a limited time in order to protect the confidentiality or proprietary nature of any information contained therein.